CLINICAL TRIAL: NCT01603823
Title: Angiographie and OCT in Macula and Retinal Diseases
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Assoc.Prof., Medical University of Vienna
Other Study IDs: 10082007
Record Dates: First submitted 2012-05-19; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Macular Edema
Keywords: vitrectomy; cataract; macular edema
MeSH Terms: conditions — Macular Edema; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy volunteers
- St.p. Pars plana vitrectomy

SUMMARY:
The purpose of this study is to investigate the morphological and angiological retinal changes in different macular diseases.

DETAILED DESCRIPTION:
Recently, a new generation of OCT devices relying on spectral domain technology (SD-OCT) has been introduced and allows for higher-resolution imaging. Based on this technology we can identify variable changes at the retinal surface such as, retinal thickening with cyst formation, swelling in the inner and outer nuclear layers and subretinal fluid. The introduction of an eye-tracking mode has allowed a better insight into the development of retinal morphologic changes The aim of this study was to investigate the incidence and structural morphology of PCME after successful uncomplicated cataract surgery in patients with previous pars plana vitrectomy (PPV) and indocyanine green-assisted peeling of an epiretinal membrane and the internal limiting membrane (ILM).

ELIGIBILITY:
Inclusion Criteria:

* previous 23-gauge PPV and ILM peeling

Exclusion Criteria:

* history of branch retinal vein occlusion
* central retinal vein occlusion
* wet macular degeneration
* diabetic retinopathy
* uveitis or other inflammatory eye disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty eyes of 20 patients with previous 23-gauge PPV and ILM peeling (PPV group) and 15 consecutive eyes with senile cataract with a healthy macula (control group) were included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Mylonas G, Sacu S, Deak G, Dunavoelgyi R, Buehl W, Georgopoulos M, Schmidt-Erfurth U; Macula Study Group Vienna. Macular edema following cataract surgery in eyes with previous 23-gauge vitrectomy and peeling of the internal limiting membrane. Am J Ophthalmol. 2013 Feb;155(2):253-259.e2. doi: 10.1016/j.ajo.2012.07.013. Epub 2012 Oct 1. PMID 23036567